CLINICAL TRIAL: NCT01082562
Title: Randomized, Double-blind, Placebo-Controlled, Ascending Single- and Multiple-Dose Study to Evaluate the Safety , Pharmacokinetics and Pharmacodynamics of BMS-844421 in Healthy Subjects and in Subjects With Elevated Cholesterol
Brief Title: Safety Study of BMS-844421 for Treatment of Hypercholesterolemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CV198-002; 2009-012032-32 (EudraCT Number)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Atherosclerosis; Hypercholesterolemia
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (16):
- Arm 1 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 2 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution
- Arm 3 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 4 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution
- Arm 5 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 6 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution
- Arm 7 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 8 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution
- Arm 9 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 10 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution
- Arm 11 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 12 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution
- Arm 13 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 14 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution
- Arm 15 - BMS-844421 (Experimental)
  Interventions: Drug: BMS-844421
- Arm 16 - 0.9% sodium chloride injection solution (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection solution

INTERVENTIONS:
Drug: BMS-844421 — Ready-to-use stock solution for SC and IV, Subcutaneous, 37.5 mg
  SAD: Once, 1 Day
  MAD: IV loading followed by 4 weekly doses, 29 Days
  Arms: Arm 1 - BMS-844421; Arm 11 - BMS-844421; Arm 13 - BMS-844421; Arm 15 - BMS-844421; Arm 3 - BMS-844421; Arm 5 - BMS-844421; Arm 7 - BMS-844421; Arm 9 - BMS-844421
Drug: 0.9% sodium chloride injection solution — Injection solution, Subcutaneous, 37.5 mg
  SAD: Once, 1 Day
  MAD: IV loading followed by 4 weekly doses, 29 Days
  Arms: Arm 10 - 0.9% sodium chloride injection solution; Arm 12 - 0.9% sodium chloride injection solution; Arm 14 - 0.9% sodium chloride injection solution; Arm 16 - 0.9% sodium chloride injection solution; Arm 2 - 0.9% sodium chloride injection solution; Arm 4 - 0.9% sodium chloride injection solution; Arm 6 - 0.9% sodium chloride injection solution; Arm 8 - 0.9% sodium chloride injection solution

SUMMARY:
The purpose of this study is to assess the safety, tolerability, serum concentrations and pharmacodynamic effects on serum low-density lipoprotein (LDL) cholesterol of single and multiple subcutaneous and intravenous doses of BMS-844421 in healthy subjects (SAD) and in subjects with elevated cholesterol (MAD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects (SAD)
* Healthy Subjects (MAD) with untreated elevated cholesterol
* Body Mass Index (BMI) of 18 to 30 kg/m² inclusive
* Women who are not of childbearing potential and men, ages 18 to 45

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of liver or renal disorders
* Prior use of any prescription or over-the-counter lipid lowering drugs, within 8 weeks prior to study drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To asses safety, tolerability, pharmacodynamic effects of BMS-844421 on PCSK9 concentrations | At the conclusion of the MAD part of the study

SECONDARY OUTCOMES:
Assess single and multiple dose pharmacokinetics of BMS-844421 | All outcomes will be assessed at the conclusion of the MAD part of the study
Assess the absolute bioavailability of single BMS-844421 SC doses | All outcomes will be assessed at the conclusion of the MAD part of the study
Assess the effects of multiple doses of BMS-844421on lipid components | All outcomes will be assessed at the conclusion of the MAD part of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Berlin, Germany

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx